CLINICAL TRIAL: NCT02817113
Title: Phase I Study of NC-6004 in Combination With 5-FU and Cetuximab as First-line Treatment in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of NC-6004 in Combination With 5-FU and Cetuximab in Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategy change
Sponsor: Orient Europharma Co., Ltd. (Industry)
Collaborators: NanoCarrier Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-006
Record Dates: First submitted 2016-06-06; First posted 2016-06-29 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — demplatin pegraglumer; Cetuximab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NC-6004, Cetuximab and 5-FU (Experimental): Cetuximab will be administered before the start of chemotherapy at a loading dose of 400 mg/m2 given, followed by a subsequent weekly doses of 250 mg/m2; NC-6004 will be administered on Day 1 every 3 weeks, and 5-FU will be administered at a dose of 1,000 mg/m2/day on Day 1- Day 4 as continuous infusion every 3 weeks.
  Interventions: Drug: NC-6004; Drug: Cetuximab; Drug: 5-FU

INTERVENTIONS:
Drug: NC-6004 — One cycle of treatment lasts for 3 weeks. NC-6004 will be administered over 1 hour on Day 1 (after the cetuximab infusion) every 3 weeks
  Other Names: Micelplatin (Taiwan only); Nanoplatin (Japan only)
Drug: Cetuximab — One cycle of treatment lasts for 3 weeks. For each cycle, cetuximab will be administered at least 1 hour before the start of chemotherapy at a loading dose of 400 mg/m2 given over 2 hours initially (ie, on the first day of treatment), followed by a subsequent weekly doses of 250 mg/m2 over 1 hour.
  Other Names: Erbitux
Drug: 5-FU — One cycle of treatment lasts for 3 weeks. 5-FU will be administered at a dose of 1,000 mg/m2/day on Day 1- Day 4 as continuous infusion every 3 weeks.
  Other Names: Fluorouracil

SUMMARY:
NC-6004 is a polymeric micelle containing cisplatin as an active moiety. The nanoparticle provides sustained release of the active moiety and utilizes the enhanced permeability and retention (EPR) effect to target release of platinum to tumors. This Phase I study aims to establish a recommended dose (RD) for the triplet combination of NC-6004 plus 5-FU and cetuximab as first-line treatment in patient with recurrent and/or metastatic squamous cell carcinoma of the head and neck for further clinical study development.

DETAILED DESCRIPTION:
1. Primary objectives

   ♦ To determine the Maximum Tolerated Dose (MTD) of NC-6004 according to the Dose Limiting Toxicity (DLT) in combination with 5-FU plus cetuximab as firstline treatment in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN), and to decide the RD for the following studies
2. Secondary objectives 1). To evaluate the safety and tolerability profile of NC-6004 in combination with 5- FU plus cetuximab 2). To assess the pharmacokinetic effects of NC-6004 3). To assess the antitumor effects of NC-6004

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Known (histology/cytology proven) or evidenced by radiology of recurrent and/or metastatic SCCHN not suited for local therapy
* Males or females aged ≥ 20 years and < 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy >12 weeks as judged by investigators
* Adequate bone marrow reservation:
* Adequate liver function:
* Adequate renal function:
* Reasonably recovered from preceding major surgery as judged by the Investigator or no major surgery within 4 weeks prior to the start of Day 1 treatment

Exclusion Criteria:

* Female of child-bearing potential who is or has intention to be pregnant or breastfeeding.
* Previous radiotherapy within 3 months before study entry
* Known brain metastasis or leptomeningeal involvement
* Marked pleural effusion or ascites above Grade 2, based on NCI-CTCAE v4.03 criteria
* History of thrombocytopenia with complications (including hemorrhage or bleeding ≥ Grade 2, based on NCI-CTCAE v4.03 criteria), hemolytic condition, or coagulation disorders that would make subjects unsafe based on the judgment of the Investigator
* Patients who have unresolved toxicity from all radiation, adjuvant/neoadjuvant chemotherapy, other targeted treatment including investigational treatment (exception of alopecia and ≤ Grade 2 peripheral neuropathy) according to NCI-CTCAE v4.03 criteria
* Known hypersensitivity to the study drugs or the drugs with similar chemical structures
* History of myocardial infarction within 6 months before study entry, unstable congestive heart failure (New York Heart Association, NYHA Stage III-IV), angina pectoris, or transient ischemic attack or cardiac arrhythmia requiring medical therapy
* History of any other cancer other than head and neck cancer (HNC) (except carcinoma in situ of the cervix) within the last 5 years.
* Primary tumor of the nasopharynx (nasopharyngeal carcinoma)
* Known HIV-1 or any active infection requiring IV antibiotics

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 29 months
  MTD of NC-6004 according to the DLT when administered in combination with 5-FU plus cetuximab as first-line treatment

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 29 months
  According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 criteria
Incidence of AE lead to treatment discontinuation | 29 months
Peak Plasma Concentration (Cmax) | Within 4 cycles (each cycle is 21 days)
Time of Maximum concentration observed (Tmax) | Within 4 cycles (each cycle is 21 days)
Area under the plasma concentration-time curve from time zero to time (AUC0-t) | Within 4 cycles (each cycle is 21 days)
Area under the concentration time-curves from time zero to infinity (AUC0-∞) | Within 4 cycles (each cycle is 21 days)
Terminal Elimination Rate Constant (λz) | Within 4 cycles (each cycle is 21 days)
Elimination Half-life (t½) | Within 4 cycles (each cycle is 21 days)
Clearance (CL) of total platinum in plasma | Within 4 cycles (each cycle is 21 days)
Clearance (CL) of total platinum in plasma ultrafiltrate | Within 4 cycles (each cycle is 21 days)
Volume of Distribution (Vz) of total platinum in plasma | Within 4 cycles (each cycle is 21 days)
Volume of Distribution (Vz) of total platinum in plasma ultrafiltrate | Within 4 cycles (each cycle is 21 days)
Tumor response rate (RR) | 29 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 on MRI or CT results
Disease control rate (DCR) | 29 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 on MRI or CT results
Overall response rate (ORR) | 29 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 on MRI or CT results

OTHER OUTCOMES:
Changes in vital signs | 29 months
  Arterial blood pressure, heart rate, respiratory rate and temperature are to be monitored during infusion.
Changes in laboratory results | 29 months
  Number of participants with abnormal laboratory values and/or adverse events that are related to treatment.
Physical examination findings | 29 months
  Number of participants with physical examination abnormal findings that are related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No